CLINICAL TRIAL: NCT01063075
Title: Phase 2 Study to Evaluate the Pharmacokinetics and Drug-Drug Interaction of Cetuximab and Carboplatin in Patients With Advanced Solid Tumors
Brief Title: A Study in Advanced Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 13420; I4E-MC-JXBB (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-02-03; First posted 2010-02-05 (Estimated); Results first posted 2016-06-15 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Solid Tumor
Keywords: Cancer of Head; Cancer of Head and Neck; Cancer of Neck; Head and Neck Cancer; Head Cancer; Head Neoplasms; Head, Neck Neoplasms; Neck Cancer; Neck Neoplasms; Solid Neoplasm; Carcinoma; Sarcoma
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma; Sarcoma | interventions — Cetuximab; Carboplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cetuximab and Carboplatin (D) (Experimental): Group D:
  Cycle 1 (1 week, combination therapy):
  400 milligrams per square meter (mg/m ²) cetuximab administered intravenously (I.V) on week 1,day 1. Carboplatin area under the curve (AUC=5) administered I.V on week 1,day 1.
  Optional 5- fluorouracil (FU) administered as a 96-hour continuous infusion (C.I.) of 1000 mg/ m ²/day administered starting on week 1, day 1.
  After 1 cycle, participants may then receive cetuximab as determined by clinical exam or radiological imaging studies until progression of disease, unacceptable toxicity, or another withdrawal criterion is met.
  After protocol amendment February 2014, any newly enrolled participants were placed into Group D only.
  Interventions: Drug: Cetuximab; Drug: Carboplatin; Drug: 5 - FU
- Cetuximab and Carboplatin (C) (Experimental): Group C: Cycle 1 (4 weeks, combination therapy): Carboplatin (AUC=5) administered I.V on week 1, day 1.1000 mg/m ²/day 5-FU administered as a 96-hour C.I. starting on week 1, day 1.
  400 mg/m² cetuximab administered I.V on week 2, day 1. 250 mg/m ² cetuximab administered I.V on week 3 and 4, day 1.
  Cycle 2-6 (3 weeks, combination therapy): Carboplatin (AUC=5) administered I.V on week1,day1.1000 mg/m ²/d 5-FU as a 96-hour C.I. starting on week1, day1. 250 mg/m ² cetuximab administered I.V on Week 1-3, day 1.
  After 6 cycles, participants may then receive cetuximab monotherapy until progression of disease, unacceptable toxicity, or another withdrawal criterion is met.Due to protocol amendment in September 2011, any newly enrolled participants were placed into cetuximab and carboplatin (C) arm only. After protocol amendment February 2014, any newly enrolled participants will be placed into Group D arm only.
  Interventions: Drug: Cetuximab; Drug: Carboplatin; Drug: 5 - FU
- Cetuximab and Carboplatin (B) (Experimental): Group B:
  Cycle 1 (3 weeks, single-agent cetuximab):
  400 mg/m² cetuximab administered I.V on week 1, day 1. 250 mg/m ² cetuximab administered I.V on weeks 2 and 3, day 1.
  Cycle 2 (3 weeks, combination therapy):
  Carboplatin (AUC=5) administered I.V week 1, day 1. 1000 mg/m ²/d 5-FU administered as a 96-hour C.I. starting on week 1, day 1. 250 mg/m ² cetuximab administered I.V weeks 1- 3,day 1.
  After 6 cycles, participants may then receive cetuximab monotherapy until progression of disease, unacceptable toxicity, or another withdrawal criterion is met.
  Due to protocol amendment in September 2011,any newly enrolled participants were placed into cetuximab and carboplatin (C) arm only. After protocol amendment February 2014, any newly enrolled participants will be placed into Group D arm only.
  Interventions: Drug: Cetuximab; Drug: Carboplatin; Drug: 5 - FU
- Carboplatin and Cetuximab (A) (Experimental): Group A:
  Cycle 1 (3 weeks, combination therapy):
  Carboplatin (AUC=5) administered I.V on week 1, day 1. 1000 mg/m ²/d 5-FU administered as a 96-hour C.I. starting on week 1, day 1.
  400 mg/m ² cetuximab administered I.V on week 2, day 1. 250 mg/m ² cetuximab administered I.V on week 3, day 1.
  Cycle 2 (3 weeks, combination therapy):
  Carboplatin (AUC=5) administered I.V on week 1, day 1. 1000 mg/m ²/d 5-FU administered as a 96-hour C.I. starting on week 1, day 1. 250 mg/m ² cetuximab administered I.V on weeks 1- 3, day 1.
  After 7 cycles, participants may then receive cetuximab monotherapy until progression of disease, unacceptable toxicity, or another withdrawal criterion is met.
  Due to protocol amendment in September 2011, any newly enrolled participants were placed into cetuximab and carboplatin (C) arm only. After protocol amendment February 2014, any newly enrolled participants will be placed into Group D arm only.
  Interventions: Drug: Cetuximab; Drug: Carboplatin; Drug: 5 - FU

INTERVENTIONS:
Drug: Cetuximab — Administered Intravenously
Drug: Carboplatin — Administered Intravenously
Drug: 5 - FU — Administered Intravenously

SUMMARY:
The primary purpose of this study is to help answer the following research question(s):

* To see how the body absorbs, processes, and gets rid of cetuximab when the drug is taken in combination with carboplatin [pharmacokinetic (PK) analysis]
* To see if any drug interactions occur between cetuximab and carboplatin.

ELIGIBILITY:
Inclusion Criteria:

* The participant has histologically or cytologically confirmed advanced solid tumor that is resistant to standard therapy or for which there is no standard therapy.
* The participant has measurable or non-measurable disease according to RECIST 1.0 guidelines.
* The participant has a life expectancy of greater than 3 months.
* The participant has an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* The participant has adequate hematologic function as defined by absolute neutrophil count greater than or equal to 1500/microliter (μL), hemoglobin greater than or equal to 9 grams/deciliter (g/dL), and platelet count greater than or equal to 100,000/μL.
* The participant has adequate hepatic function as defined by a total bilirubin less than or equal to 2 x the upper limit of normal (ULN), aspartate transaminase (AST, SGOT) and alanine transaminase (ALT, SGPT) less than or equal to 3 x the ULN (or less than or equal to 5 x the ULN in the presence of known liver metastases).
* The participant has adequate renal function as defined by serum creatinine less than or equal to 1.5 x the institutional ULN or creatinine clearance greater than or equal to 60 mL/min for participants with creatinine levels above the ULN.
* The participant has the ability to understand, and the willingness to sign, a written informed consent document.
* If the participant has received prior therapy with platinum, the time to the first treatment of study drug from the last platinum exposure is >28 days.

Exclusion Criteria:

* The participant has symptomatic brain or leptomeningeal metastasis.
* The participant has not recovered from adverse events due to agents administered more than 4 weeks earlier. Neurotoxicity, if present, must have improved to Grade less than 2 per the National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) v 3.0.
* The participant is receiving any other investigational agent(s).
* The participant is receiving concurrent treatment with other anticancer therapy, including chemotherapy, immunotherapy, hormonal therapy,radiation therapy ( RT), chemoembolization, or targeted therapy. Participants receiving palliative radiation therapy to bony metastases prior to the first dose of study medication are eligible.
* The participant is receiving therapy with immunosuppressive agents.
* The participant has known drug or alcohol abuse.
* The participant has uncontrolled hypertension defined as systolic blood pressure greater than or equal to 180 millimeters of mercury (mm Hg) or diastolic blood pressure greater than or equal to 130 mm Hg.
* The participant has a history of allergic reactions attributed to compounds of chemical or biologic composition similar to those of cetuximab or carboplatin.
* The participant has a medical or psychological condition that would not permit the participant to complete the study or sign informed consent.
* The participant has clinically relevant coronary artery disease or history of myocardial infarction in the last 12 months or high risk of uncontrolled arrhythmia or uncontrolled cardiac insufficiency.
* The participant, if female, is pregnant (confirmed by serum or urine beta-human chorionic gonadotropin [β-HCG] pregnancy test) or breastfeeding
* The participant has had a known positive test result for the human immunodeficiency virus.
* The participant has an active infection (requiring I.V antibiotics), including tuberculosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-06; Primary Completion 2015-05 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST, Study Director — Eli Lilly and Company
Locations (8):
- United States (6):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - University of Kansas Medical Center, Fairway, Kansas
  - Portland VA Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Canada (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to protocol amendment in September 2011, any newly enrolled participants were placed into cetuximab and carboplatin (C) arm only. After protocol amendment February 2014, any newly enrolled participants were placed into Group D arm only.
Groups:
- Carboplatin and Cetuximab (A): Group A:
  Cycle 1 (3 weeks, combination therapy):
  Carboplatin (AUC=5) administered I.V on week 1, day 1. 1000 mg/m ²/d 5-FU administered as a 96-hour C.I. starting on week 1, day 1.
  400 milligrams per square meter (mg/m ²) cetuximab administered I.V on week 2, day 1. 250 mg/m ² cetuximab administered I.V on week 3, day 1.
  Cycle 2 (3 weeks, combination therapy):
  Carboplatin (AUC=5) administered I.V on week 1, day 1. 1000 mg/m ²/d 5-FU administered as a 96-hour C.I. starting on week 1, day 1. 250 mg/m ² cetuximab administered I.V on weeks 1- 3, day 1.
- Cetuximab and Carboplatin (B): Group B:
  Cycle 1 (3 weeks, single-agent cetuximab):
  400 mg/m² cetuximab administered I.V on week 1, day 1. 250 mg/m ² cetuximab administered I.V on weeks 2 and 3, day 1.
  Cycle 2 (3 weeks, combination therapy):
  Carboplatin (AUC=5) administered I.V week 1, day 1. 1000 mg/m ²/d 5-FU administered as a 96-hour C.I. starting on week 1, day 1. 250 mg/m ² cetuximab administered I.V weeks 1- 3,day 1.
- Cetuximab and Carboplatin (C): Group C:
  Cycle 1 (4 weeks, combination therapy):
  Carboplatin (AUC=5) administered I.V on week 1, day 1.1000 mg/m ²/day 5-FU administered as a 96-hour C.I. starting on week 1, day 1.
  400 mg/m² cetuximab administered I.V on week 2, day 1. 250 mg/m ² cetuximab administered I.V on week 3 and 4, day 1.
  Cycle 2-6 (3 weeks, combination therapy):
  Carboplatin (AUC=5) administered I.V on week1,day1.1000 mg/m ²/d 5-FU as a 96-hour C.I. starting on week1, day1. 250 mg/m ² cetuximab administered I.V on Week 1-3, day 1.
- Cetuximab and Carboplatin (D): Cycle 1 (1 week, combination therapy):
  400 milligrams per square meter (mg/m ²) cetuximab administered intravenously (I.V) on week 1, day 1. Carboplatin area under the curve (AUC=5) administered I.V on week 1, day 1.
  Optional 5- fluorouracil (FU) administered as a 96-hour continuous infusion (C.I.) of 1000 mg/ m ²/day administered starting on week 1, day 1.
Period: Overall Study
Arm/Group | Carboplatin and Cetuximab (A) | Cetuximab and Carboplatin (B) | Cetuximab and Carboplatin (C) | Cetuximab and Carboplatin (D)
Started | 2 | 3 | 14 | 15
Completed | 1 | 1 | 9 | 14
Not Completed | 1 | 2 | 5 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- All Participants (Group A, B, C and D): Group D:
  Cycle 1:400 mg/m² cetuximab week (w) 1,day(d) 1.Carboplatin(AUC=5) on w 1, d 1.Optional 1000 mg/m²/d 5-FU given as a 96-hour C.I. starting(strt) on w 1, d 1.
  Group C:
  Cycle 1:Carboplatin(AUC=5) on w 1,d 1. 400 mg/m² cetuximab on w 2, d 1.Cetuximab 250 mg/m ² on w 3 and 4, d 1.
  Cycle 2-6:Carboplatin(AUC=5) and 250 mg/m² cetuximab on w 1, d 1.1000 mg/m²/d 5-FU given as a 96-hour C.I. strt on w 1, d 1.250 mg/m² cetuximab on w 2 and 3, d 1.
  Group B:
  Cycle 1:400 mg/m² cetuximab on w 1, d 1. 250 mg/m ² cetuximab on w 2 and 3, d 1.
  Cycle 2:Carboplatin(AUC=5) w 1, d 1.1000 mg/m ²/d 5-FU given as 96-hour C.I. strt on w 1, d 1. 250 mg/m ² cetuximab w 1- 3, d 1.
  Group A:
  Cycle 1:Carboplatin(AUC=5) on w 1, d 1. 1000 mg/m²/d 5-FU given as 96-hour C.I. strt on w 1, d 1.
  400 mg/m² cetuximab on w 2, d 1 and 250 mg/m² cetuximab on w 3, d 1. Cycle 2:Carboplatin(AUC=5) given I.V on w 1, d 1.1000 mg/m²/d 5-FU given as 96-hour C.I. strt on w 1, d 1. 250 mg/m² cetuximab on w 1-3, d 1.
Arm/Group | All Participants (Group A, B, C and D)
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.20 (12.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 31
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Canada | 10
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Total Carboplatin Pharmacokinetics (PK): Area Under the Concentration (AUC) Versus Time Curve From Time Zero to Infinity (AUC[0-∞])
Time Frame: Group D: Cycle 1, Week 1, Day 1; Prior to Carboplatin Infusion, 1hour (H), 1:30 H, 2 H, 3 H, 5 H, 8 H, 24 H, 72 H (after the Start of Carboplatin Infusion)
Population: Participants who received at least 1 dose of study drug who were enrolled in Group(Grp)D & had evaluable PK data.Study design by intent did not collect data from Grp B.Due to participant recruitment & retention challenges,there were no PK study completers for Grp A & C.Participant recruitment & retention addressed by amending protocol to add Grp D.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hour/milliliters (μg•h/mL)
Groups:
- Cetuximab and Carboplatin (D): Group D:
  Cycle 1 (1 week, combination therapy):
  400 milligrams per square meter (mg/m ²) cetuximab administered intravenously (I.V) on week 1, day 1. Carboplatin area under the curve (AUC=5) administered I.V on week 1, day 1.
  Optional 5- fluorouracil (FU) administered as a 96-hour continuous infusion (C.I.) of 1000 mg/ m ²/day administered starting on week 1, day 1.
Arm/Group | Cetuximab and Carboplatin (D)
Number analyzed (Participants) | 13
micrograms*hour/milliliters (μg•h/mL) | 129 (14.8)

2. Primary Outcome: Cetuximab PK: Area Under the Concentration Versus Time Curve During One Dosing Interval at Steady State (AUC τ,ss)
Time Frame: (Group B: Cycle 1 and Cycle 2+ ; Day 1, 8, 15 and Group C: Cycle 1, Day 8, 15 and 22; Cycle 2+, Day 1,8 and 15): Prior to Cetuximab Infusion, 1 Hour (H), 2 H, 4 H, 8 H, 24 H, 72 H, 120 H, and 168 H (after the start of Cetuximab Infusion)
Population: All participants who received at least one dose of study drug who were enrolled in Group B and C and had evaluable PK data. Study design by intent did not collect data from Groups D and A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hour/milliliters (μg•h/mL)
Groups:
- Cetuximab (B and C); Cetuximab and Carboplatin (B and C): Group B:
  Cycle 1 (3 weeks, single-agent cetuximab):
  400 mg/m² cetuximab administered I.V on week 1, day 1. 250 mg/m ² cetuximab administered I.V on weeks 2 and 3, day 1.
  Cycle 2 (3 weeks, combination therapy):
  Carboplatin (AUC=5) administered I.V week 1, day 1. 1000 mg/m ²/d 5-FU administered as a 96-hour C.I. starting on week 1, day 1. 250 mg/m ² cetuximab administered I.V weeks 1- 3,day 1.
  Group C:
  Cycle 1 (4 weeks, combination therapy):
  Carboplatin (AUC=5) administered I.V on week 1, day 1.1000 mg/m ²/day 5-FU administered as a 96-hour C.I. starting on week 1, day 1.
  400 mg/m² cetuximab administered I.V on week 2, day 1. 250 mg/m ² cetuximab administered I.V on week 3 and 4, day 1.
  Cycle 2-6 (3 weeks, combination therapy):
  Carboplatin (AUC=5) administered I.V on week1,day1.1000 mg/m ²/d 5-FU as a 96-hour C.I. starting on week1, day1. 250 mg/m ² cetuximab administered I.V on Week 1-3, day 1.
Arm/Group | Cetuximab (B and C) | Cetuximab and Carboplatin (B and C)
Number analyzed (Participants) | 5 | 5
micrograms*hour/milliliters (μg•h/mL) | 17200 (15.8) | 16700 (18.5)

3. Primary Outcome: Total Carboplatin PK: Maximum Observed Plasma Concentration (Cmax)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliters (μg/mL)
Arm/Group | Cetuximab and Carboplatin (D)
Number analyzed (Participants) | 13
micrograms per milliliters (μg/mL) | 11.5 (15.8)

4. Primary Outcome: Cetuximab PK: Maximum Observed Plasma Concentration at Steady State (Cmax,ss)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliters (μg/mL)
Arm/Group | Cetuximab (B and C) | Cetuximab and Carboplatin (B and C)
Number analyzed (Participants) | 5 | 5
micrograms per milliliters (μg/mL) | 199 (10.3) | 199 (10.8)

5. Primary Outcome: Total Carboplatin PK: Time of Maximum Observed Plasma Concentration (Tmax)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | Cetuximab and Carboplatin (D)
Number analyzed (Participants) | 13
Hour (h) | 1.12 [1.00 to 1.30]

6. Primary Outcome: Cetuximab PK: Time of Maximum Observed Plasma Concentration at Steady State (Tmax,ss)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | Cetuximab (B and C) | Cetuximab and Carboplatin (B and C)
Number analyzed (Participants) | 5 | 5
Hour (h) | 1.15 [1.02 to 7.83] | 3.17 [2.00 to 4.07]

7. Primary Outcome: Cetuximab PK: Confirmatory Serum Concentration
Time Frame: Group D: Prior to Carboplatin Infusion, Cycle 1, Day 1
Population: All participants who received at least one dose of study drug who were enrolled in Group D and had evaluable PK data. Study design by intent did not collect data from Groups A, B, and C.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliters (µg/mL)
Groups:
- Cetuximab (D): Group D:
  Cycle 1 (1 week, combination therapy):
  400 milligrams per square meter (mg/m ²) cetuximab administered intravenously (I.V) on week 1, day 1. Carboplatin area under the curve (AUC=5) administered I.V on week 1, day 1.
  Optional 5- fluorouracil (FU) administered as a 96-hour continuous infusion (C.I.) of 1000 mg/ m ²/day administered starting on week 1, day 1.
Arm/Group | Cetuximab (D)
Number analyzed (Participants) | 14
micrograms per milliliters (µg/mL) | 195 (16.5)

ADVERSE EVENTS:
Groups:
- Carboplatin and Cetuximab (A): Group A:
  Cycle 1 (3 weeks, combination therapy):
  Carboplatin (AUC=5) administered I.V on week 1, day 1. 1000 mg/m ²/d 5-FU administered as a 96-hour C.I. starting on week 1, day 1.
  400 mg/m ² cetuximab administered I.V on week 2, day 1. 250 mg/m ² cetuximab administered I.V on week 3, day 1.
  Cycle 2 (3 weeks, combination therapy):
  Carboplatin (AUC=5) administered I.V on week 1, day 1. 1000 mg/m ²/d 5-FU administered as a 96-hour C.I. starting on week 1, day 1. 250 mg/m ² cetuximab administered I.V on weeks 1- 3, day 1.
- Carboplatin and Cetuximab (B): Group B:
  Cycle 1 (3 weeks, single-agent cetuximab):
  400 mg/m² cetuximab administered I.V on week 1, day 1. 250 mg/m ² cetuximab administered I.V on weeks 2 and 3, day 1.
  Cycle 2 (3 weeks, combination therapy):
  Carboplatin (AUC=5) administered I.V week 1, day 1. 1000 mg/m ²/d 5-FU administered as a 96-hour C.I. starting on week 1, day 1. 250 mg/m ² cetuximab administered I.V weeks 1- 3,day 1.
- Carboplatin and Cetuximab (C): Group C:
  Cycle 1 (4 weeks, combination therapy):
  Carboplatin (AUC=5) administered I.V on week 1, day 1.1000 mg/m ²/day 5-FU administered as a 96-hour C.I. starting on week 1, day 1.
  400 mg/m² cetuximab administered I.V on week 2, day 1. 250 mg/m ² cetuximab administered I.V on week 3 and 4, day1.
  Cycle 2-6 (3 weeks, combination therapy):
  Carboplatin (AUC=5) administered I.V on week1,day1.1000 mg/m ²/d 5-FU as a 96-hour C.I. starting on week1, day1. 250 mg/m ² cetuximab administered I.V on Week 1-3, day 1.
- Carboplatin and Cetuximab (D): Group D:
  Cycle 1 (1 week, combination therapy):
  400 milligrams per square meter (mg/m ²) cetuximab administered intravenously (I.V) on day 1. Carboplatin area under the curve (AUC=5) administered I.V on day 1.
  Optional 5- fluorouracil (FU) administered as a 96-hour continuous infusion (C.I.) of 1000 mg/ m ²/day administered starting on day 1.
Arm/Group | Carboplatin and Cetuximab (A) | Carboplatin and Cetuximab (B) | Carboplatin and Cetuximab (C) | Carboplatin and Cetuximab (D)
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/3 | 5/14 | 10/15
Other Adverse Events (participants affected / at risk) | 2/2 | 2/3 | 14/14 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin and Cetuximab (A) (N=2) | Carboplatin and Cetuximab (B) (N=3) | Carboplatin and Cetuximab (C) (N=14) | Carboplatin and Cetuximab (D) (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Obstructive uropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal haematoma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Carboplatin and Cetuximab (A) (N=2) | Carboplatin and Cetuximab (B) (N=3) | Carboplatin and Cetuximab (C) (N=14) | Carboplatin and Cetuximab (D) (N=15)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 4 (6) | 6 (15)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (8) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (9) | 3 (5)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 3 (3)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (3) | 5 (5) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 8 (14) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 7 (9) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (4) | 11 (25) | 8 (10)
Salivary gland disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 5 (8) | 4 (5)
Tongue haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (11) | 6 (14) | 5 (5)
Asthenia (General disorders) | 1 (1) | 0 (0) | 4 (6) | 1 (1)
Catheter site bruise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site rash (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased activity (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (9) | 7 (10) | 9 (11)
Infusion site rash (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Local swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 1 (1) | 7 (23) | 3 (4)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 3 (4) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Opportunistic infection (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeding tube complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Human bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Alanine aminotransferase decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breath sounds abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 2 (6) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Monocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (2) | 2 (2) | 1 (3)
Platelet count decreased (Investigations) | 1 (4) | 1 (3) | 3 (4) | 6 (20)
Weight decreased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (11) | 5 (6)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 4 (7) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3) | 9 (13)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (9) | 6 (11)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (3) | 3 (7)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Magnesium deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 3 (5) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 3 (4)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle tone disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Reflexes abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 4 (5) | 1 (1)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1/4 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1/4 (1)
Vulvovaginal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1/4 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (5) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 7 (15) | 9 (14)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hirsutism (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1/4 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (11) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (6) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to protocol amendment in September 2011, any newly enrolled participants were placed into cetuximab and carboplatin(C) arm only. After protocol amendment February 2014, any newly enrolled participants were placed into Group D arm only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days